CLINICAL TRIAL: NCT07207382
Title: Clinical and Radiographic Evaluation of Three Biomimetic Materials in Pulp Therapy of Immature Young Permanent Teeth "A Randomized Controlled Clinical Trial"
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Mohamed Fakhry, phd candidate of pediatric dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED23-5D
Record Dates: First submitted 2025-10-02; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Pulpotomy of Young Permanent Molars
Keywords: young permanent; MTA; Pulpotomy; premixed bioceramic; treated dentin matrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: MTA group
- B (Experimental)
  Interventions: Drug: Premixed Bioceramic material
- C (Experimental)
  Interventions: Drug: Treated Dentin Matrix

INTERVENTIONS:
Drug: MTA group — MTA group is considered the control group
  Arms: A
Drug: Premixed Bioceramic material — Premixed Bioceramic material is test group B
  Arms: B
Drug: Treated Dentin Matrix — Treated Dentin Matrix is test group C
  Arms: C

SUMMARY:
Statement of the problem:

Pulpotomy is the most popular technique for maintaining vitality and has a substantial impact on continuing root growth in vital, young permanent molars suffering from dental cavities.

Biomimetic materials placement after performing pulp therapy is one of the important factors to determine healing of the pulp and continue root formation. In this study a novel material "Treated Dentin Matrix" is used in comparison to premixed bioceramic material and "Mineral Trioxide Aggregate" in pulpotomy of immature permanent molars.

The Aim of the study:

Is to assess the clinical and radiographic success of pulpotomized first permanent immature molars treated with three different Biomimetic materials (Treated Dentin Matrix, Premixed Bio-ceramic material and Mineral Trioxide Aggregate)

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 7 and 10 years-old.
2. Vital permanent first molars with deep caries lesion approaches the pulp without symptoms of irreversible pulpitis, with open apices in the radiograph.
3. Permanent first molars with pulpal exposure that occurred during caries excavation.
4. Incompletely formed roots

Exclusion Criteria:

* (1) Teeth with signs and symptoms of chronic infection such as swelling and mobility. (2) Teeth with excessive bleeding from amputated radicular stumps (3) Teeth showing radiographic evidence of pathologic root resorption, inter-radicular bone loss, periapical pathology and calcifications in the canals. (4) Lack of patient/parent compliance and cooperation. (5)Children who are physically or mentally disabled or having any medical condition that will complicate the treatment

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 18 months
  * Absence of pain related to the treated teeth, Including patient reported pain or sensitivity to percussion/palpation.
  * No evidence of swelling of supporting soft tissue or presence of sinus tract.
  * Absence of excessive mobility affecting treated teeth.
Radiographic success | 18 months
  * Radiographic criteria for success in terms of:
  * Progression of root formation
  * No Internal or external root resorption.
  * No Periapical or furcal radiolucency.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No